CLINICAL TRIAL: NCT00112905
Title: Phase II Trial of Sorafenib (BAY 43-9006) (IND 69896; NSC 724772) in Patients With Advanced Urothelial Cancer
Brief Title: Sorafenib in Treating Patients With Regional or Metastatic Cancer of the Urothelium
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02975; NCI-2012-02975 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA021115 (NIH); E1804 (Other: Eastern Cooperative Oncology Group); E1804 (Other: CTEP)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2011-04-04 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2012-12

CONDITIONS: Adenocarcinoma of the Bladder; Distal Urethral Cancer; Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Proximal Urethral Cancer; Recurrent Bladder Cancer; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Urethral Cancer; Regional Transitional Cell Cancer of the Renal Pelvis and Ureter; Squamous Cell Carcinoma of the Bladder; Stage III Bladder Cancer; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder; Urethral Cancer Associated With Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-56. Courses repeat every 56 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with progressive regional or metastatic cancer of the urothelium. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the 4-month progression-free survival rate, response rate and toxicity of BAY 43-9006 in patients with progressing regional or metastatic transitional cell carcinoma (or mixed histologies containing a component of TCC) of the urothelium who have progressed on one and only one prior systemic chemotherapy regimen for metastatic disease.

SECONDARY OBJECTIVES:

I. To determine the time to disease progression and overall survival with BAY 43-9006.

II. To evaluate the frequency of polymorphisms in drug metabolizing enzymes and to correlate these polymorphisms with variations in BAY 43-9006 pharmacokinetics.

III. To evaluate the frequency of raf kinase mutations in tumor specimens and correlate these with response rate.

IV. To evaluate serum VEGF levels as potential markers of angiogenesis inhibition by BAY 43-9006.

V. To evaluate markers of apoptosis and kinase inhibition in peripheral blood mononuclear cells as potential biomarkers of BAY 43-9006 activity.

VI. To determine if there are proteins differentially translated from the genome in patients who respond to treatment with BAY 43-9006 versus patients who do not respond to BAY 43-9006.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-56. Courses repeat every 56 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months until 2 years from study entry and then every 6 months until 3 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed transitional cell carcinoma or mixed histologies containing a component of transitional cell carcinoma of the urothelium (renal pelvis, ureter, bladder, urethra) with manifestations of progressing regional or metastatic cancer; or (2) Nontransitional cell histologies include patients with adenocarcinoma or squamous cell carcinomas representing greater than 90% of specimen; patients with small cell carcinoma, soft tissue sarcomas, or carcinosarcomas are excluded
* Measurable disease, as defined in the RECIST criteria; all sites of disease must be evaluated within 4 weeks prior to registration
* Patients must have progressed on one and only one prior systemic chemotherapy for metastatic disease; prior chemotherapy administered in the adjuvant or neoadjuvant setting is permitted (i.e. does not count as 1 prior regimen) provided that it was completed greater than 12 months prior to the start of the first chemotherapy regimen administered in the metastatic setting
* Patients must not have had prior systemic biologic response modifier therapy; patients must not have had chemotherapy, hormonal or biologic therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or have recovered from adverse events due to agents administered more than 4 weeks earlier
* Prior radiotherapy is allowed; patients must be >= 2 weeks post-radiotherapy at time of registration; a previously irradiated lesion can only be used as a marker lesion if there is unequivocal evidence of progression demonstrated on serial imaging studies; patients must have recovered from all toxicities associated with prior radiotherapy
* Patients must be >= 4 weeks post-major surgery at time of registration; patients must have recovered from all toxicities associated with prior surgery
* ECOG performance status of 0 or 1
* No history of severe cardiovascular disease (AHA Class III or IV), uncontrolled CHF, uncontrolled hypertension, or ventricular dysrhythmias
* Patients with previously resected and irradiated CNS metastases with evidence of stable disease are eligible
* Patients with a history of prior malignancy are eligible provided they were treated with curative intent and have been disease free for >= 5 years; curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the cervix must have been treated with curative intent; patients with clinically unsuspected organ confined prostate cancer found at the time of cystoprostatectomy are eligible
* Creatinine < 1.5 mg/dL
* Granulocytes >= 1500/mm^3
* Platelets >= 100,000/mm^3
* AST =< 2.5 x institutional upper limit of normal
* Bilirubin < 1.5 mg/dl
* No active unresolved infection requiring parenteral antibiotics < 7 days prior to study entry
* Patients must not have a swallowing dysfunction which would prevent the ingesting of pills
* Patients must not have any evidence of bleeding diathesis
* Patients must not be on therapeutic anticoagulation; prophylactic anticoagulation (i.e. low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for PT, INR or PTT are met
* Patients must not be taking the cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine, and phenobarbital), rifampin, or St. John's Wort
* Women of childbearing potential must not be pregnant (as proven by a negative pregnancy test within 14 days prior to registration) or breast feeding because the effects of this treatment on the fetus and breast-fed infants is unknown
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreicer, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 10/26/2005. The TCC (transitional cell carcinoma) cohort was suspended for an efficacy evaluation on 10/30/2006 after reaching its first stage accrual goal. A total of 27 patients entered the TCC cohort, and no patient entered the non-TCC cohort. The study was terminated on March 10th, 2008.
Groups:
- TCC (Transitional Cell Carcinoma) Cohort: Sorafenib was administered at a dose of 400 mg orally twice daily (total daily dose 800 mg) for eight weeks as one cycle. Patients swallowed the tablets whole with approximately 250 ml (8 oz.) of water each morning and evening (i.e., 12-hourly), with or without food. If sorafenib was taken with meals, patients were instructed to take sorafenib tosylate with a moderate to low-fat meal, as a high fat meal caused a decrease in absorption in previous studies. Patients were instructed to keep a pill diary and record the pills they took each day.
Period: Overall Study
Arm/Group | TCC (Transitional Cell Carcinoma) Cohort
Started | 27
Eligible and Treated | 22
Completed | 15
Not Completed | 12
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Ineligibility | 5
Not completed — Alternative treatment | 1
Not completed — performance status was deteiorating | 1

BASELINE CHARACTERISTICS:
Groups:
- TCC Cohort: Only eligible and treated patients are included in the analysis.
  BAY 43-9006 was administered at a dose of 400 mg orally twice daily (total daily dose 800 mg) for eight weeks as one cycle. Patients swallowed the tablets whole with approximately 250 ml (8 oz.) of water each morning and evening (i.e., 12-hourly), with or without food. If Bay 43-9006 was taken with meals, patients were instructed to take BAY 43-9006 tosylate with a moderate to low-fat meal, as a high fat meal caused a decrease in absorption in previous studies.
Arm/Group | TCC Cohort
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 66 [37 to 81]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of eligible participants who began treatment.
  Participants
    Female | 8
    Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Progression-free Survival at 4 Months
Description: Survival estimate from the Kaplan-Meier curve of the proportion of patients alive and progression-free at 4 months.
  Progression-free survival is defined as the time from registration to progression or death, whichever occurs first.
  Progression is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s) or unequivocal progression of existing nontarget lesions.
Time Frame: Assessed every cycle while on treatment; after being off-treatment, assessed every 3 months for 2 years, then every 6 months for 1 year.
Population: Per protocol, the primary analysis included eligible patients who started protocol treatment.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | TCC Cohort
Number analyzed (Participants) | 22
Percentage of Participants | 11 [0 to 23]

2. Secondary Outcome: Progression-free Survival
Description: Time from registration to the earlier of disease progression or death. Patients alive and progression-free at last follow-up were censored.
  Progression is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s) or unequivocal progression of existing nontarget lesions.
Time Frame: as for outcome 1
Population: Only eligible and treated patients are included in this analysis.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | TCC Cohort
Number analyzed (Participants) | 22
Months | 2.2 [1.8 to 3.7]

3. Secondary Outcome: Overall Survival
Description: Time from registration to death. Patients alive at last follow-up were censored.
Time Frame: as for outcome 1
Population: Only eligible and treated patients are included in this analysis.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | TCC Cohort
Number analyzed (Participants) | 22
Months | 6.8 [5.7 to 8.5]

4. Secondary Outcome: Best Overall Response by RECIST
Description: This outcome measure reports the best response a patient has ever experienced.
  <Target Lesions>
  Complete Response (CR):
  The disappearance of all target lesions, confirmed by assessments >=4 weeks (wks) later.
  Partial Response:
  >=30% decrease in the sum of the longest diameters of target lesions from baseline, confirmed by assessments >=4 wks later.
  Progressive Disease (PD):
  >=20% increase in the sum of the longest diameters of target lesions from the smallest sum longest diameter since baseline, or the appearance of new lesions.
  Stable Disease (SD):
  Neither response criteria nor progressive disease criteria are met for >=8 wks.
  <Nontarget Lesions>
  CR:
  The disappearance of all nontarget lesions and normalization of tumor marker levels, confirmed by assessments >=4 wks later.
  SD:
  Persistence of nontarget lesions or maintenance of tumor marker levels above the normal limits for >=8 wks.
  PD:
  The appearance of new lesions or unequivocal progression of existing lesions.
Time Frame: as for outcome 1
Population: Only eligible and treated patients are included in the analysis.
Measure: Number; unit: Participants
Arm/Group | TCC Cohort
Number analyzed (Participants) | 22
Participants
  Complete response | 0
  Partial response | 0
  Stable disease | 3
  Progression | 9
  Unevaluable | 10

ADVERSE EVENTS:
Time Frame: Assessed every 8 weeks
Arm/Group | TCC Cohort
Serious Adverse Events (participants affected / at risk) | 15/27
Other Adverse Events (participants affected / at risk) | 24/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TCC Cohort (N=27)
Hypertension (Vascular disorders) | 1
Fatique (General disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 5
Hyperthyroidism, thyrotoxicosis (Endocrine disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TCC Cohort (N=27)
Hypertension (Vascular disorders) | 8
Fatigue (General disorders) | 14
Weight loss (Investigations) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 10
Constipation (Gastrointestinal disorders) | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 7
Mucositis/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 9
Taste disturbance (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
ALT increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less